CLINICAL TRIAL: NCT01759459
Title: A Comparison of Lidocaine, Buffered Lidocaine, and Bacteriostatic Normal Saline for Local Anesthesia Prior to Peripheral Intravenous Catheterization
Brief Title: Local Anesthetics for Pain Reduction Prior to IV Line Placement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, David Gurda, Principal Investigator/PharmD, Allina Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3867-1
Record Dates: First submitted 2012-12-27; First posted 2013-01-03 (Estimated); Results first posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Pain; Local Anesthesia for Peripheral Intravenous Catheterization
MeSH Terms: conditions — Pain | interventions — Lidocaine; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lidocaine (Experimental): 1% Lidocaine for injection, 0.50 mL administered one time intradermally in peripheral forearm
  Interventions: Drug: Lidocaine
- Buffered Lidocaine (Experimental): 1% Buffered Lidocaine for injection, 0.50 mL administered one time intradermally in peripheral forearm
  Buffered lidocaine is compounded by the following process:
  2.3 mLs of 8.4% sodium bicarbonate is added to a vial of 1% lidocaine
  Interventions: Drug: Buffered Lidocaine
- Bacteriostatic Normal Saline (Experimental): Bacteriostatic Normal Saline for injection, 0.50 mL administered one time intradermally in peripheral forearm
  Interventions: Drug: Bacteriostatic Normal Saline

INTERVENTIONS:
Drug: Lidocaine — The medication will be administered immediately prior to receiving peripheral IV catheter placement
  Other Names: Hospira brand 1% Lidocaine in 20 mL vial
  Arms: Lidocaine
Drug: Buffered Lidocaine — The medication will be administered immediately prior to receiving peripheral IV catheter placement
  Other Names: Hospira brand 1% Lidocaine in 20 mL vial; Hospira brand 8.4% sodium bicarbonate in 50 mL vial
  Arms: Buffered Lidocaine
Drug: Bacteriostatic Normal Saline — The medication will be administered immediately prior to receiving peripheral IV catheter placement
  Other Names: Hospira brand Bacteriostatic Normal Saline in 10 mL vial
  Arms: Bacteriostatic Normal Saline

SUMMARY:
The purpose of this study is to compare the pain level felt by patients when receiving placement of a peripheral intravenous catheter (IV line) following the administration of a local anesthetic. The local anesthetics tested will be lidocaine, buffered lidocaine, and bacteriostatic normal saline. Lidocaine is commonly used as a premedication for reducing the pain upon insertion of peripheral IV lines. However, due to its acidic nature, the lidocaine itself may cause pain upon administration. To help counter this discomfort, pharmacies can "buffer" the lidocaine using sodium bicarbonate, which increases the pH to a neutral value, resulting in less pain. Bacteriostatic normal saline has also been used for local anesthesia with peripheral IV placement, particularly in patients with a lidocaine allergy, as it contains benzyl alcohol which acts as a local anesthetic.

There are minimal reports from the literature that directly compare patient reported pain of all three agents to one another, although studies do exist that have compared buffered lidocaine versus lidocaine and buffered lidocaine versus bacteriostatic normal saline. To address this comparison gap, the following research questions need to be asked: which anesthetic agent is the superior premedication for reducing the amount of pain upon administration of the local anesthetic itself and for the pain associated with the peripheral insertion of the catheter? The hypothesis of the investigators is that there is not a significant difference in the degree of pain scales between the anesthetic agents to justify the pharmacoeconomic costs associated with compounding buffered lidocaine.

The primary outcome measured in this study will be the level of pain reported by the patient upon administration of the local anesthetic and upon insertion of the peripheral intravenous catheter. A secondary outcome includes a pharmacoeconomic analysis that will look specifically at the cost-savings of using one agent over the other and will take into account the daily time allocated to pharmacy technicians and pharmacists for compounding and verifying buffered lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 18 y.o.
* Ability to speak, read, an/or understand English
* Ability to communicate a level of pain via the specified pain scale
* A written order exists for an intravenous peripheral catheter insertion for the patient

Exclusion Criteria:

* Lidocaine allergy
* Buffered lidocaine allergy
* Benzyl alcohol allergy
* Non-English speaking
* Non-responsive or unable to understand or report pain score (ex. intubated in the ICU)
* Inability to place catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Gurda, PharmD, Principal Investigator — Allina Health Services
Locations (1):
- United Hospital, part of Allina Health Services, Saint Paul, Minnesota, United States

REFERENCES:
- [Result] Beck RM, Zbierajewski FJ, Barber MK, Engoren M, Thomas R. A comparison of the pain perceived during intravenous catheter insertion after injection with various local anesthetics. AANA J. 2011 Aug;79(4 Suppl):S58-61. PMID 22403968
- [Result] Brown D. Local anesthesia for vein cannulation: a comparison of two solutions. J Infus Nurs. 2004 Mar-Apr;27(2):85-8. doi: 10.1097/00129804-200403000-00004. PMID 15085035
- [Result] Carvalho B, Fuller A, Brummel C, Cohen SE. Local infiltration of epinephrine-containing lidocaine with bicarbonate reduces superficial bleeding and pain during labor epidural catheter insertion: a randomized trial. Int J Obstet Anesth. 2007 Apr;16(2):116-21. doi: 10.1016/j.ijoa.2006.09.006. Epub 2007 Feb 5. PMID 17276670
- [Result] Cornelius P, Kendall J, Meek S, Rajan R. Alkalinisation of lignocaine to reduce the pain of digital nerve blockade. J Accid Emerg Med. 1996 Sep;13(5):339-40. doi: 10.1136/emj.13.5.339. PMID 8894861
- [Result] Burke SD, Vercler SJ, Bye RO, Desmond PC, Rees YW. Local anesthesia before IV catheterization. Am J Nurs. 2011 Feb;111(2):40-5; quiz 46-7. doi: 10.1097/01.NAJ.0000394291.40330.3c. PMID 21270583
- [Result] Fatovich DM, Jacobs IG. A randomized controlled trial of buffered lidocaine for local anesthetic infiltration in children and adults with simple lacerations. J Emerg Med. 1999 Mar-Apr;17(2):223-8. doi: 10.1016/s0736-4679(98)00157-7. PMID 10195475
- [Result] Ganter-Ritz V, Speroni KG, Atherton M. A randomized double-blind study comparing intradermal anesthetic tolerability, efficacy, and cost-effectiveness of lidocaine, buffered lidocaine, and bacteriostatic normal saline for peripheral intravenous insertion. J Infus Nurs. 2012 Mar-Apr;35(2):93-9. doi: 10.1097/NAN.0b013e31824241cc. PMID 22382793
- [Result] McNaughton C, Zhou C, Robert L, Storrow A, Kennedy R. A randomized, crossover comparison of injected buffered lidocaine, lidocaine cream, and no analgesia for peripheral intravenous cannula insertion. Ann Emerg Med. 2009 Aug;54(2):214-20. doi: 10.1016/j.annemergmed.2008.12.025. Epub 2009 Feb 13. PMID 19217695
- [Result] Nakayama M, Munemura Y, Kanaya N, Tsuchida H, Namiki A. Efficacy of alkalinized lidocaine for reducing pain on intravenous and epidural catheterization. J Anesth. 2001;15(4):201-3. doi: 10.1007/s005400170003. PMID 14569436
- [Result] Windle PE, Kwan ML, Warwick H, Sibayan A, Espiritu C, Vergara J. Comparison of bacteriostatic normal saline and lidocaine used as intradermal anesthesia for the placement of intravenous lines. J Perianesth Nurs. 2006 Aug;21(4):251-8. doi: 10.1016/j.jopan.2006.05.007. PMID 16935736

RESULTS

PARTICIPANT FLOW:
Groups:
- Buffered Lidocaine: 1% Buffered Lidocaine for injection, 0.50 mL administered one time intradermally in peripheral forearm
  Buffered lidocaine is compounded by the following process:
  2.3 mLs of 8.4% sodium bicarbonate is added to a vial of 1% lidocaine
  Buffered Lidocaine: The medication will be administered immediately prior to receiving peripheral IV catheter placement
Period: Overall Study
Arm/Group | Lidocaine | Buffered Lidocaine | Bacteriostatic Normal Saline
Started | 50 | 50 | 50
Completed | 50 | 50 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Buffered Lidocaine | Bacteriostatic Normal Saline | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Mean (Full Range); unit: years] | 58.3 [20 to 75] | 56.6 [20 to 75] | 56 [20 to 75] | 57.5 [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 29 | 78
  Male | 26 | 25 | 21 | 72
Baseline pain scores [Mean (Full Range); unit: units on a scale] — The outcome measured will be the level of pain reported, on a scale of 0 to 10, 0 being no pain at all and 10 being the worst pain ever felt, by the patient upon administration of the local anesthetic and upon insertion of the peripheral intravenous catheter. Baseline pain scores were also recorded using this same scale
  units on a scale | 0.09 [0 to 10] | 0.03 [0 to 10] | 0.15 [0 to 10] | 0.09 [0 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Following Anesthetic Administration
Description: The primary outcome measured in this study will be the level of pain reported, on a scale of 0 to 10, 0 being no pain at all and 10 being the worst pain ever felt, by the patient upon administration of the local anesthetic and upon insertion of the peripheral intravenous catheter.
Time Frame: Day 1
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lidocaine | Buffered Lidocaine | Bacteriostatic Normal Saline
Number analyzed (Participants) | 50 | 50 | 50
units on a scale | 2.81 [0 to 10] | 1.64 [0 to 10] | 2.05 [0 to 10]

2. Secondary Outcome: Economic Analysis of Cost of Compounding Buffered Lidocaine Versus Cost of Purchasing Regular Lidocaine and/or Bacteriostatic Normal Saline
Description: A secondary outcome includes a pharmacoeconomic analysis that will look specifically at the cost-savings of using one agent over the other and will take into account the daily time allocated to pharmacy technicians and pharmacists for compounding and verifying buffered lidocaine. The outcome data was measured and reported in a single value dollar amount per group, tallied over a 3 month period. The dollar amounts were estimated by adding up the costs of drug purchasing, technician compounding time, and pharmacist verifying time. Buffered lidocaine required both drug purchasing and compounding time, where the lidocaine and bacteriostatic normal saline required drug purchasing alone and labor costs were not taken into account.
Time Frame: 3 months
Population: An analysis adding up the costs of drug purchasing, technician compounding time, and pharmacist verifying time, within a quarter of a year. Buffered lidocaine required both drug purchasing and compounding time, where the lidocaine and bacteriostatic normal saline required drug purchasing alone and labor costs were not taken into account.
Measure: Number; unit: Dollars
Units Other Than Participants: Medication vials
Groups:
- Buffered Lidocaine Cost: An analysis adding up the costs of drug purchasing, technician compounding time, and pharmacist verifying time. Based on salaries during this period, technician costs = $0.03/minute and pharmacist costs = $1.00/minute.
- Lidocaine Cost; Bacteriostatic Normal Saline Cost: An analysis adding up the costs of drug purchasing alone.
Arm/Group | Buffered Lidocaine Cost | Lidocaine Cost | Bacteriostatic Normal Saline Cost
Number analyzed (Participants) | 50 | 50 | 50
Number analyzed (Medication vials) | 9676 | 9676 | 9676
Dollars | 13400 | 9100 | 4840

3. Other Pre Specified Outcome: Pain Score Following Peripheral Catheter Insertion
Description: as for outcome 1
Time Frame: Baseline and day 1
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lidocaine | Buffered Lidocaine | Bacteriostatic Normal Saline
Number analyzed (Participants) | 50 | 50 | 50
units on a scale
  Average pain score following medication injection | 2.58 [0 to 10] | 1.6 [0 to 10] | 2.10 [0 to 10]
  Average pain score following IV inserti | 1.81 [0 to 10] | 1.81 [0 to 10] | 3.05 [0 to 10]

ADVERSE EVENTS:
Arm/Group | Lidocaine | Buffered Lidocaine | Bacteriostatic Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No